CLINICAL TRIAL: NCT07367971
Title: Open-Label, Within-Subject Drug-Drug Interaction Study of ABP-671 Added to Stable Allopurinol Therapy in Gout Patients
Brief Title: Drug-Drug Interaction Study of ABP-671 in Gout Patients
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Atom Therapeutics Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABP-671-DDI-01
Record Dates: First submitted 2025-12-27; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-12

CONDITIONS: Gout Chronic; Gout; DDI (Drug-Drug Interaction)
Keywords: gout; Gout Chronic; ABP-671
MeSH Terms: conditions — Gout | interventions — Allopurinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ABP-671 (Experimental)
  Interventions: Drug: ABP-671 plus allopurinol

INTERVENTIONS:
Drug: ABP-671 plus allopurinol — All subjects undergo three sequential 7-day periods:
  Period 1 (Day 1-7): Allopurinol；
  Period 2 (Day 1-7): Allopurinol Plus ABP-671；
  Period 3 (Day 1-7): ABP-671；

SUMMARY:
This is a open-Label, Within-Subject Drug-Drug Interaction Study of ABP-671 Added to Stable Allopurinol Therapy in Gout Patients. Pharmacokinetic (PK) interaction between ABP-671 and Allopurinol will be evaluated in participants who are on stable Allopurinol therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-75 years with clinical diagnosis of gout.
* Stable Allopurinol therapy QD for ≥14 days prior to Day 1.
* Cohort N: Normal renal function.
* Cohort R: Moderate renal impairment.

Exclusion Criteria:

* Clinically significant hepatic impairment.
* History of Allopurinol hypersensitivity.
* Pregnancy or breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-26 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of allopurinol | Base line, through Day1, Day 7,Day8,D14,D15,D21
  Maximum observed plasma concentration (Cmax) of allopurinol following administration of allopurinol alone and in combination with ABP-671 at steady state.
Area under the plasma concentration-time curve over the dosing interval (AUC) of allopurinol | Base line, through Day1, Day 7,Day8,D14,D15,D21
  Area under the plasma concentration-time curve over the dosing interval (AUC) of allopurinol following administration of allopurinol alone and in combination with ABP-671 at steady state.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of ABP-671 | Though Day7,Day8,Day14,Day15,Day21
  Maximum observed plasma concentration (Cmax) of ABP-671 when administered with allopurinol and following a post-combination ABP-671 alone period.
Area under the plasma concentration-time curve over the dosing interval (AUC) of ABP-671 | Though Day7,Day8,Day14,Day15,Day21
  Area under the plasma concentration-time curve over the dosing interval (AUC) of ABP-671 when administered with allopurinol and following a post-combination ABP-671 alone period.
Incidence of treatment-emergent adverse events (TEAEs) | Through study completion, an average of 51 days
  Number and percentage of participants experiencing treatment-emergent adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Wakefield Clinical Research, Cary, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
there is no need at present.